CLINICAL TRIAL: NCT05621954
Title: Telehealth for Pre- and Post-Operative Monitoring of Cardiac Surgery Patients - A Randomised Controlled Trial
Brief Title: Telehealth Interventions for Cardiac Surgery
Acronym: TICS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Liverpool Heart and Chest Hospital NHS Foundation Trust (Other)
Collaborators: Liverpool Centre for Cardiovascular Science (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: TICS
Record Dates: First submitted 2022-10-25; First posted 2022-11-18 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-05

CONDITIONS: Cardiac Valve Disease; Coronary Artery Disease; Surgical Complication
Keywords: Telehealth; Remote Monitoring; Waiting List; Quality of Life
MeSH Terms: conditions — Heart Valve Diseases; Coronary Artery Disease | interventions — Remote Patient Monitoring

STUDY DESIGN:
Intervention Model Description: Pragmatic, single-centre, individual patient, randomized controlled trial
Masking Description: No masking
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telehealth monitoring (Experimental): Telehealth remote monitoring provided by a specialised service with a monitoring and patient education app featuring:
  * Symptom, blood pressure, weight, heart rate and oxygen saturation monitoring with optional step counters
  * Customised algorithms with patient feedback for prehabilitation (e.g. patient self-reporting of symptoms, activities and health-related activities with positive feedback loops and recommendations for self-directed management)
  * Centralised weekly review and escalation to expedited surgery if deteriorations noted
  * Post-operative monitoring with symptom, blood pressure, weight, heart rate, oxygen saturation and photographic wound review with optional step counters
  Interventions: Procedure: Telehealth Monitoring
- Standard of Care (No Intervention): Standard of care will be no remote monitoring for patients whilst on the waiting list or after discharge from hospital. Access to tertiary services for advice, information or to report deteriorations will be through conventional existing modes such as printed or online literature provided at the time of outpatient review, telephone access to administrative staff allowing clinical information to be conveyed to the usual care team, and local primary care and emergency services for acute deteriorations. Existing standard of care remote services (e.g. wound monitoring by digital photograph reviews) will continue.

INTERVENTIONS:
Procedure: Telehealth Monitoring — Connected devices and smartphone apps to measure symptoms and observations at home, with centralisation of results to a staffed hub
  Other Names: Docobo; Remote Monitoring; Doc@Home
  Arms: Telehealth monitoring

SUMMARY:
The goal of this clinical trial is to compare telehealth monitoring at home against usual care in patients undergoing planned heart surgery. The main questions it aims to answer are:

1. Can telehealth improve quality of life prior to surgery
2. Can telehealth prevent serious deterioration requiring hospital or primary care attendance

Participants awaiting heart surgery will be randomly allocated to either telehealth remote monitoring of symptoms, blood pressure, heart rate, oxygen levels and activity levels or they will be allocated to usual care which is unmonitored on the waiting list for surgery.

Researchers will compare telehealth to usual care to see if it improves quality of life or prevents deteriorations on the waiting list.

DETAILED DESCRIPTION:
Patients on elective cardiac surgery waiting lists can deteriorate, presenting via acute services as urgent inpatients as a result of their decompensation and facing increased surgical risk. With increases in waiting times prevalent through the country, and healthcare resources under pressure from Covid-related backlogs, it is imperative to find ways to monitor and escalate the most vulnerable patients and to provide safe methods of providing healthcare interventions outside conventional hospital settings. Remote monitoring identifies patients at need, and allows tertiary-care led interventions to prevent deterioration in the first instance. Such facilities could also enhance recovery following treatment and reduce the risks of complications and readmissions post-operatively.

The benefits and risks of such programmes is, however, not well understood: additional monitoring may increase the burden of responsibility on patients or monitoring facilities without providing additional safeguards to the patient. The advantages of early detection may not translate into improved outcomes and the onus on the patient to report in may reduce quality of life rather than enhance it.

The researchers therefore seek to identify if telehealth monitoring can improve health related quality of life, reduce unplanned admissions and healthcare resource utilisation and enhance pre-habilitation using protocolised patient engagement facilities to reduce complications and improve risk-stratification metrics such as smoking status, diabetic control and BMI.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients over 18y referred and accepted for cardiac surgery
2. Able to consent to participate

Exclusion Criteria:

1. Urgent or emergent surgery
2. Surgery planned within 3 weeks of first cardiac surgery outpatient review

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 318 (Actual)
Dates: Start 2023-04-04 (Actual); Primary Completion 2025-08-08 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Change from baseline to admission in Healthcare related Quality of Life Change (EQ5D5L) | From baseline to admission for surgery (up to 52 weeks)
  EQ5D5L will be measured by electronic questionnaire by the patient or a researcher on their behalf and indexed for representation on a scale from 0 (worst health, equivalent to being dead) - 1 (best health). The difference in measures between baseline (randomisation) and admission for surgery (up to 52 weeks) will be measured.
Healthcare resource use during waiting list (composite counts of admission to hospital, A&E attendance and primary care appointment utilisation) | From baseline (randomisation) to admission for surgery (up to 52 weeks)
  Composite counts of admissions to hospital, Accident & Emergency hospital attendance, and primary care appointments for this health condition or complications of this health condition adjudicated by the research team. The counts will be accrued from baseline (randomisation) to admission for surgery (up to 52 weeks).

SECONDARY OUTCOMES:
Unplanned admissions pre- and post-surgery | From baseline to discharge from outpatient cardiac surgery service (up to 52 weeks)
  Rates of unplanned admissions to hospital both pre- and post- surgery
Diabetes control | From baseline (randomisation) to admission for surgery (up to 52 weeks)
  Change from baseline to admission on HbA1c
Smoking cessation | From baseline (randomisation) to admission for surgery (up to 52 weeks)
  Change from baseline to admission on HbA1c
Post-operative Quality of Life Measures | From discharge from hospital admission to discharge from outpatient cardiac surgery service (up to 52 weeks)
  Healthcare related Quality of Life Change (EQ5D5L change) as an indexed measure from 0 (worst health, equivalent to being dead) to 1 (best health).
Change in post-operative complications | From discharge from hospital admission to discharge from outpatient cardiac surgery service (up to 52 weeks)
  Rates of post-operative complications including mortality, stroke, lower respiratory tract infections, surgical site infections
Length of hospital stay | From admission for surgery to discharge from hospital (up to 52 weeks)
  Total in-hospital stay
Ventilator Time | From admission for surgery to discharge from hospital (up to 52 weeks)
  Total cumulative time with invasive ventilation following index procedure
Length of intensive care stay | From admission for surgery to discharge from hospital (up to 52 weeks)
  Total critical care stay for index admission
Weight loss | From baseline (randomisation) to admission for surgery (up to 52 weeks)
  Change in body mass index on waiting list

CONTACTS AND LOCATIONS:
Locations (1):
- Liverpool Heart and Chest Hospital, Liverpool, Mersey, United Kingdom

IPD SHARING:
Plan to Share IPD: No
There is no plan to make data widely available. However, should a legitimate request be made by bona fide researchers with data protection legislation equivalent to European Union or United Kingdom General Data Protection Regulations (GDPR), this would not be discounted out of hand. Governance procedures to fully anonymise all identifiable details would be required for any individual participant data, but protocols, analytic source code, data collection forms etc would be shared after publication of the study.